CLINICAL TRIAL: NCT03569813
Title: Making it Last: A Randomized, Controlled Trial of a Home Care System to Promote Persistence in PrEP Care
Brief Title: Pre-exposure Prophylaxis (PrEP) at Home
Acronym: PrEP@Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Aaron Siegler, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00096594; R01MH114692 (NIH)
Record Dates: First submitted 2018-06-15; First posted 2018-06-26 (Actual); Results first posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: HIV/AIDS
Keywords: Pre-exposure prophylaxis (PrEP); Home-based monitoring
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: This trial will include 396 participants with 2:1 allocation for the intervention (264) and control (132) conditions. The sample of 396 will target inclusion of 50% Black and 50% younger (aged 18-34) participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PrEP@Home System (Experimental): The experimental group will be assigned to the remote care system for one year of follow-up PrEP care to include home test kits, behavioral surveillance, and telemedicine visits as needed.
  Interventions: Behavioral: PrEP@Home System
- Standard of Care (Active Comparator): The comparator group will receive active linkage to a local PrEP provider for clinic-based PrEP follow-up. Participants in this study arm will be seen quarterly by a health care provider, per standard of care when taking PrEP.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Behavioral: PrEP@Home System — The PrEP@Home system includes a home care kit mailed quarterly to participants. The kit has components for self-collection of urine, rectal and pharyngeal swabs, microtube blood collection, and materials for return shipping. Biological tests routinely performed at PrEP follow-up (FU) visits will be done on the specimens. At months 6 and 12, the kit will include materials to assess for protective levels of emtricitabine triphosphate (FTC-TP).
  The system includes a study app through which participants may track the mailing of home testing kits, access quarterly surveys, and communicate with study clinicians. The surveys will include domains that physicians assess at PrEP care quarterly FU visits (sexual risk, illicit substance use, PrEP adherence, side effects).
  Study Clinicians will review Lab and survey results and if the results show no contraindications for PrEP continuation, the clinician may renew a participant's PrEP prescription. Telemedicine visits will be scheduled as needed.
  Arms: PrEP@Home System
Other: Standard of Care — Control participants will receive clinic-based PrEP follow-up. After the baseline assessment, control participants will receive active linkage to standard, clinic-based PrEP care for their next PrEP care follow-up visit. Participants will also download the control version of the study app, which will contain only research elements pertinent to their participation in the control arm of the study including quarterly surveys. At months 6 and 12, control arm participants will be sent materials for DBS self-collection and return shipping to allow for measurement of the study outcome, emtricitabine triphosphate (FTC-TP).
  Arms: Standard of Care

SUMMARY:
This study is a randomized clinical trial of PrEP@Home, a home care system for Human Immunodeficiency Virus (HIV) Pre-Exposure Prophylaxis (PrEP). Individuals entering into PrEP care at an initial in-person study visit will be randomized to the PrEP@Home system for home-based PrEP care follow-up visits or to the control standard of care for clinic-based follow-up visits. The primary aim of this study is to assess protective levels of PrEP medication for the intervention arm compared to the control arm.

DETAILED DESCRIPTION:
Clinical guidance calls for quarterly follow-up visits for individuals taking PrEP. Yet these visits impose burdens on the healthcare system and on patients that could hinder the persistence of patients in PrEP care. Preliminary data indicate that a home-based care system for PrEP is feasible, and acceptable, and may increase patient willingness to remain in care.

This study explores the effect of a home-based PrEP support system on maintenance in PrEP care. The study will enroll 396 participants in a stratified randomized, controlled trial comparing the PrEP@Home intervention arm to the standard of care control arm. The study seeks to explore intervention performance among highly impacted groups and therefore will target a sample that is 50% Black and 50% aged 18-34 years.

Individuals in the intervention and control arms will have a baseline study visit, in which patients will be prescribed PrEP. Participants randomized to the intervention arm will receive home care for PrEP at months 3, 6, 9, and 12. Home care will include a mailed package with materials for HIV/sexually transmitted infection (STI)/creatinine specimen self-collection, materials for return shipping, and a link to an electronic, self-report behavioral assessment. Home care will also include access to the intervention version of the study app to facilitate patient-provider and patient-system interactions. Study clinicians will monitor participants' in-home care, and renew prescriptions as indicated. Control arm participants will be linked to a local PrEP provider, where they will be seen for quarterly clinic visits per standard of care. Control participants will have access to the control version of the study app that contains only research elements pertinent to their participation in the control arm of the study.

ELIGIBILITY:
Inclusion Criteria:

* Male at birth
* Report anal sex with a man in the past 6 months
* Are able to complete survey instruments in English
* Live in the metropolitan area of a study site
* Are willing to provide at least 2 means of alternate contact
* Willing to not enroll in another HIV prevention trial
* HIV-negative (self-reported and lab confirmed)
* Own and willing to use a smartphone for the duration of the study
* Willing to download the study app
* Willing to take a photo of a PrEP prescription label
* Behaviorally indicated for PrEP (per Centers for Disease Control and Prevention (CDC) guidance) or African American men who have sex with men (MSM) who report anal sex in the last six months
* PrEP naïve or < 3 months lifetime experience of PrEP use or stopped taking PrEP >6 months ago
* Willing to take PrEP, including adherence to daily dosing
* Willing to use, as needed, study-provided PrEP navigation services to obtain coverage for PrEP medication
* Able to work with the study site to develop a plan to cover the financial cost of PrEP if not covered through insurance or Gilead financial assistance
* Willing to use a home kit that will include a self-administered collection of urine, rectal and pharyngeal swabs, and finger prick blood.

Exclusion Criteria:

* Reports having genital reassignment surgery
* <18 or ≥ 50 years of age
* Currently enrolled in another HIV prevention trial
* Symptoms of acute HIV infection, or being evaluated for acute infection because of recent high-risk exposure
* Currently taking PEP
* Creatinine clearance <60 ml/min
* Contraindications to taking tenofovir disoproxil fumarate/emtricitabine (TDF/FTC) or tenofovir alafenamide/emtricitabine (TAF/FTC)
* History of hemophilia
* Unable to conduct finger prick at a study site
* Multiple screening attempts

Ages: 18 Years to 49 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 318 (Actual)
Dates: Start 2019-04-26 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2023-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Siegler, PhD, Principal Investigator — Emory University; Kenneth Mayer, MD, Principal Investigator — Harvard Medical School (HMS and HSDM)
Locations (5):
- United States (5):
  - Emory University, PRISM Health, Atlanta, Georgia
  - The Fenway Institute, Boston, Massachusetts
  - Open Arms Health Care Center, Jackson, Mississippi
  - Washington University AIDS Clinical Trial Unit, St Louis, Missouri
  - MetroHealth, Cleveland, Ohio

REFERENCES:
- [Derived] Gonzalez J, Rebolledo PA, Siegler AJ, Huang W, Mayer KH, Cantos VD. Development of a home-based pre-exposure prophylaxis care delivery system for long-acting injectable cabotegravir: a formative exploration of patient preferences. AIDS Care. 2024 Dec;36(12):1882-1890. doi: 10.1080/09540121.2024.2397128. Epub 2024 Sep 8. PMID 39245031

RESULTS

PARTICIPANT FLOW:
Recruitment Details: PrEP@Home study participants were recruited predominantly online in the study cities of Atlanta, GA, Boston, MA, Cleveland, OH, Jackson, MS, and St. Louis, MO. Participant enrollment began April 26, 2019, and all follow-up was complete by April 15, 2023. Study completion is defined as enrolled persons completing their online survey.
Groups:
- PrEP@Home System: The experimental group will be assigned to the remote care system for one year of follow-up PrEP care to include home test kits, behavioral surveillance, and telemedicine visits as needed.
  PrEP@Home System: The PrEP@Home system includes a home care kit mailed quarterly to participants. The kit has components for self-collection of urine, rectal and pharyngeal swabs, microtube blood collection, and materials for return shipping. Biological tests routinely performed at PrEP follow-up (FU) visits will be done on the specimens. At months 6 and 12, the kit will include materials to assess for protective levels of emtricitabine triphosphate (FTC-TP).
  The system includes a study app through which participants may track the mailing of home testing kits, access quarterly surveys, and communicate with study clinicians. The surveys will include domains that physicians assess at PrEP care quarterly FU visits (sexual risk, illicit substance use, PrEP adherence, side effects).
  Study Clinicians will review Lab and survey results and if the results show no contraindications for PrEP continuation, the clinician may renew a participant's PrEP prescription. Telemedicine visits will be scheduled as needed.
Period: Overall Study
Arm/Group | PrEP@Home System | Standard of Care
Started | 211 | 107
Completed | 126 | 62
Not Completed | 85 | 45

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PrEP@Home System | Standard of Care | Total
Number analyzed (Participants) | 211 | 107 | 318
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.12 (7.16) | 29.31 (7.38) | 29.58 (7.30)
Age, Customized [Count of Participants; unit: Participants]
  Between 18-24 years | 63 | 27 | 90
  Between 25-34 years | 105 | 57 | 162
  Between 35-44 years | 29 | 17 | 46
  Between 45-49 years | 14 | 6 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 211 | 107 | 318
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 15 | 33
  Not Hispanic or Latino | 192 | 89 | 281
  Unknown or Not Reported | 1 | 3 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Native Hawaiian or Pacific Islander/Asian | 6 | 6 | 12
  Black or African American | 69 | 29 | 98
  White | 119 | 53 | 172
  More than one race | 11 | 9 | 20
  Unknown or not reported | 4 | 9 | 13
Region of Enrollment [Number; unit: participants]
  United States | 211 | 107 | 318

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving Appropriate Levels of Tenofovir-diphosphate (TFV-DP) at 6-month Follow-up
Description: Adherence to study medications was measured using blood TFV-DP levels. For participants taking emtricitabine/tenofovir disoproxil fumarate, TFV-DP levels >1000 femtomole per blood spot (fmol/punch) indicated adherence of >4 doses per week. For those taking emtricitabine/tenofovir alafenamide, TFV-DP levels >140 femtomole per blood spot (fmol/punch) indicated adherence of >4 doses per week. Participants achieving these levels were considered to have adhered appropriately (>4 doses per week). Researchers used decision rules to determine adherence for participants who either reported using both medications in the period or did not report which medication they used. For instance, if a participant had a TFV-DP level above both cut points, they would be considered adherent to treatment.
Time Frame: Month 6
Population: This analysis includes participants who submitted a dry blood spot card that had an adequate size of the blood sample for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | PrEP@Home System | Standard of Care
Number analyzed (Participants) | 113 | 63
Participants | 78 | 39

2. Secondary Outcome: Retention in PrEP Care
Description: Retention in PrEP care is based on participant self-report of taking PrEP at least 4 days per week in the last week as measured at the 6 months.
Time Frame: Up to Month 6
Population: Participants with self-report data indicating adherent daily PrEP dosing.
Measure: Count of Participants; unit: Participants
Arm/Group | PrEP@Home System | Standard of Care
Number analyzed (Participants) | 155 | 77
Participants | 132 | 55

3. Secondary Outcome: Number of Participants Achieving Appropriate Levels of Tenofovir-diphosphate (TFV-DP) at 12-month Follow-up
Description: Adherence to study medications was measured using blood TFV-DP levels. For participants taking emtricitabine/tenofovir disoproxil fumarate, TFV-DP levels >1000 femtomole per blood spot (fmol/punch) indicated adherence >4 doses per week. For those taking emtricitabine/tenofovir alafenamide, TFV-DP levels >140 femtomole per blood spot (fmol/punch) indicated adherence >4 doses per week. Participants achieving these levels were considered to have adhered appropriately (>4 doses per week). For participants who either reported using both medications in the period or did not report which medication they used, the researchers used decision rules to determine adherence. For instance, if a participant had a TDF-DP level above both cutpoints, they would be considered adherent to treatment.
Time Frame: Month 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | PrEP@Home System | Standard of Care
Number analyzed (Participants) | 86 | 56
Participants | 56 | 36

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected beginning at the time consent to participate in the study was given, during study participation up to 12 months
Arm/Group | PrEP@Home System | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/211 | 0/107
Serious Adverse Events (participants affected / at risk) | 0/211 | 0/107
Other Adverse Events (participants affected / at risk) | 7/211 | 1/107
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PrEP@Home System (N=211) | Standard of Care (N=107)
STI (Infections and infestations) | 3 (3) | 0 (0)
Traveler's diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Exacerbation of Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Fracture of Ankle (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rash (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-08-08): https://cdn.clinicaltrials.gov/large-docs/13/NCT03569813/Prot_SAP_001.pdf
  • Informed Consent Form (2023-02-22): https://cdn.clinicaltrials.gov/large-docs/13/NCT03569813/ICF_002.pdf